CLINICAL TRIAL: NCT00826709
Title: CLINICAL STUDY PROTOCOL for the Prospective Evaluation of the fluID Rapid Influenza Test
Brief Title: Prospective Evaluation of the Fluid Rapid Influenza Test
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The 2008-09 North American peak influenza season ended prior to study completion.
Sponsor: Nanogen, Inc. (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Philip Estes/Associate Director, Clinical, Nanogen, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLU-05
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): 2 Nasal swabs
  Interventions: Device: fluID Rapid Influenza Test
- Arm 2 (Experimental): 2 Nasopharyngeal swabs
  Interventions: Device: fluID Rapid Influenza Test
- Arm 3 (Experimental): Nasal wash or aspirate
  Interventions: Device: fluID Rapid Influenza Test

INTERVENTIONS:
Device: fluID Rapid Influenza Test — The fluID™ Rapid Influenza Test is an in vitro diagnostic assay designed to be used with a reader for the qualitative detection of influenza type A and type B nucleoprotein antigens, and the differentiation of influenza type A subtypes A/H1 and A/H3 antigens associated with the seasonal influenza H1N1 and H3N2, in nasal swabs, nasopharyngeal swabs and nasal wash/aspirate specimens. The test is intended as an aid in the rapid, qualitative diagnosis of influenza type A and type B viral infections in patients symptomatic with influenza-like illness. The fluID™ Rapid Influenza Test is intended for use by a healthcare professional in a laboratory or Point-of-Care (POC).

SUMMARY:
The primary objective of this study is to evaluate the fluID Rapid Influenza Test's ability in detecting influenza A and influenza B from individuals presenting with signs and symptoms of influenza-like illness (ILI).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the clinical sensitivity and specificity of the fluID Rapid Influenza Test in detecting influenza A and influenza B, as evaluated with respect to fresh samples collected prospectively from individuals presenting with signs and symptoms of influenza-like illness (ILI). Test results will be compared with those obtained from viral culture testing of samples using the same specimen types, obtained from the same subjects. The specimen types under evaluation in this study will be nasal swab, nasopharyngeal swab, nasal wash and aspirate specimens.

A secondary objective of this study is to evaluate the accuracy of the fluID Rapid Influenza Test in detecting each of the H1 and H3 subtypes of influenza A, in nasal swab, nasopharyngeal swab, nasal wash and aspirate specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of any age;
2. Subjects presenting to the investigative site within 4 days of symptom onset, with:

   * Fever ≥ 38.0°C (100.4°F) if taken orally, or ≥ 38.5°C (101.2°F) if taken rectally; or a self-reported history of fever or feeling feverish (includes fever controlled by medication) in the absence of documented fever;
   * One or more respiratory symptoms of influenza-like illness which may include the following:
   * Sore throat;
   * Runny or stuffy nose;
   * Cough;
   * One or more constitutional symptoms of influenza-like illness which may include the following:
   * Myalgia (aches and pains);
   * Headache;
   * Fatigue;
3. Subjects (or parent/guardian) willing and able to provide informed consent. Written subject informed consent for this study protocol must be obtained prior to study enrollment. Each subject (or parent or guardian) must personally sign and date the Subject Informed Consent Form prior to his/her participation in this clinical study.

Exclusion Criteria:

1. Subjects not presenting with at least three symptoms of influenza-like illness as outlined above.
2. Subjects who have received influenza antiviral medication or an investigational influenza drug treatment within the previous 30 days of study enrollment.
3. Subjects (children and adults) for whom the obtaining of swab samples, nasal wash or aspirate samples is contraindicated or not possible.
4. Subjects with a medical condition that prevents swab samples or nasal washes or aspirate samples from being obtained.
5. Active duty military personnel (participating military study sites only).
6. Subjects (or parent/guardian) unwilling or unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of influenza A and influenza B | End of study

SECONDARY OUTCOMES:
Sensitivity and specificity of influenza A subtypes H1N1 and H3N2 | End of study

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - Naval Health Research Center, San Diego, California
  - University Clinical Research - DeLand, LLC, DeLand, Florida
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - The Family Doctor Research, Shreveport, Louisiana
  - Sinai Grace Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University at St. Louis, St Louis, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Granger Medical Clinic, West Valley City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University of Hong Kong, Hong Kong, Hong Kong